CLINICAL TRIAL: NCT06768957
Title: Qualitative and Quantitative Analysis of the "Single Hop Test" Combined With a Cognitive Task, to Optimize Return to Sport After Anterior Cruciate Ligament Reconstruction.
Brief Title: Test of Return to Sport After ACL Reconstruction and Cognitive Task.
Acronym: AQQSHTATC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon VALOT (Other)
Responsible Party: Sponsor-Investigator, Simon VALOT, Principal Investigator, Étudiant
Organization: Étudiant (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-A02038-39
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: ACL Reconstruction; Cognitive Function; Single Leg Hop Firm Surface; Testing Effect of Intervention

STUDY DESIGN:
Intervention Model Description: Two groups are present in parallel:
  * A control group (healthy volunteers).
  * A test group (patients who have undergone ACL reconstruction).
  Several sub-groups are present within these groups in order to carry out a crossover study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Control group: SLHD then SLHD with cognitive task (Experimental): This control group, made up of healthy subjects, will perform a single leg hop for distance and then one week later will perform a single leg hop for distance plus a cognitive task.
  Intervention 1 administered : Other: Single leg hop for distance. Intervention 2 administered : Other: Single leg hop for distance plus cognitive task.
  Interventions: Other: Single leg hop for distance; Other: Single leg hop for distance plus cognitive task
- Control group: SLHD with cognitive task then SLHD (Experimental): This control group, made up of healthy subjects, will perform a single leg hop for distance plus a cognitive task and then one week later will perform a single leg hop for distance.
  Intervention 1 administered : Other: Single leg hop for distance plus cognitive task Intervention 2 administered : Other: Single leg hop for distance
  Interventions: Other: Single leg hop for distance; Other: Single leg hop for distance plus cognitive task
- Control group: SLHD then SLHD (Experimental): This control group, made up of healthy subjects, will perform a single leg hop for distance and then one week later will perform another single leg hop for distance.
  Intervention 1 administered : Other: Single leg hop for distance Intervention 2 administered : Other: Single leg hop for distance
  Interventions: Other: Single leg hop for distance
- Control group: SLHD with cognitive task then SLHD with cognitive task (Experimental): This control group, made up of healthy subjects, will perform a single leg hop for distance plus a cognitive task and then one week later will perform another single leg hop for distance plus a cognitive task.
  Intervention 1 administered : Other: Single leg hop for distance plus cognitive task Intervention 2 administered : Other: Single leg hop for distance plus cognitive task
  Interventions: Other: Single leg hop for distance plus cognitive task
- Test group: SLHD then SLHD with cognitive task (Experimental): This test group, made up of patients who have undergone ACL reconstruction, will perform a single leg hop for distance and then one week later will perform a single leg hop for distance plus a cognitive task.
  Intervention 1 administered : Other: Single leg hop for distance. Intervention 2 administered : Other: Single leg hop for distance plus cognitive task.
  Interventions: Other: Single leg hop for distance; Other: Single leg hop for distance plus cognitive task
- Test group: SLHD with cognitive task then SLHD (Experimental): This test group, made up of patients who have undergone ACL reconstruction, will perform a single leg hop for distance plus a cognitive task and then one week later will perform a single leg hop for distance.
  Intervention 1 administered : Other: Single leg hop for distance plus cognitive task Intervention 2 administered : Other: Single leg hop for distance
  Interventions: Other: Single leg hop for distance; Other: Single leg hop for distance plus cognitive task
- Test group: SLHD then SLHD (Experimental): This test group, made up of patients who have undergone ACL reconstruction, will perform a single leg hop for distance and then one week later will perform another single leg hop for distance.
  Intervention 1 administered : Other: Single leg hop for distance Intervention 2 administered : Other: Single leg hop for distance
  Interventions: Other: Single leg hop for distance
- Test group: SLHD with cognitive task then SLHD with cognitive task (Experimental): This test group, made up of patients who have undergone ACL reconstruction, will perform a single leg hop for distance plus a cognitive task and then one week later will perform another single leg hop for distance plus a cognitive task.
  Intervention 1 administered : Other: Single leg hop for distance plus cognitive task Intervention 2 administered : Other: Single leg hop for distance plus cognitive task
  Interventions: Other: Single leg hop for distance plus cognitive task

INTERVENTIONS:
Other: Single leg hop for distance — Patients will have to perform a Single leg hop for distance.
  A 10-minute warm-up is required beforehand, followed by three single-leg hop round trips over a distance of 6m to ensure that they are able to perform the exercise.
  You start on the healthy side to understand the principles and reassure yourself. The distance covered is measured. This tells us something about the strength of the lower limb. The landing should be assessed qualitatively.
  1. Patient balanced on 1 foot, hands crossed over shoulders. 2. Jump as far as possible.
  3. Stabilise 1 time, keeping hands on shoulders.
  Arms: Control group: SLHD then SLHD; Control group: SLHD then SLHD with cognitive task; Control group: SLHD with cognitive task then SLHD; Test group: SLHD then SLHD; Test group: SLHD then SLHD with cognitive task; Test group: SLHD with cognitive task then SLHD
Other: Single leg hop for distance plus cognitive task — Patients were asked to perform a single leg hop for distance in addition to a cognitive task.
  A 10-minute warm-up is required beforehand, followed by three single-leg hop round trips over a distance of 6m to ensure that they are able to perform the exercise.
  You start on the healthy side to understand the principles and reassure yourself. The distance covered is measured. This tells us something about the strength of the lower limb. The landing should be assessed qualitatively.
  1. Patient balanced on 1 foot, hands crossed over shoulders.
  2. Observe a sequence of 5 digits, appearing every 4 seconds, on the computer in front of you.
  3. As soon as the 5th digit appears, jump as far as you can.
  4. Stabilise 1 time, keeping your hands on your shoulders.
  5. Replay the sequence of 5 numbers that appear on the screen, in reverse order.
  Arms: Control group: SLHD then SLHD with cognitive task; Control group: SLHD with cognitive task then SLHD; Control group: SLHD with cognitive task then SLHD with cognitive task; Test group: SLHD then SLHD with cognitive task; Test group: SLHD with cognitive task then SLHD; Test group: SLHD with cognitive task then SLHD with cognitive task

SUMMARY:
After reconstruction of the anterior cruciate ligament, the aim for the vast majority of sportspeople is to return to the field. To date, 65% of patients who have undergone ACL rehabilitation return to their previous level, and 55% return to competition. To achieve this, physiotherapy sessions need to prepare the return to sport as well as possible, by simulating the cognitive demands (reading the game, double task, etc.) that might be encountered on the pitch. Tests to assess the athlete's performance do exist, in order to optimise this return to sport, but they do not include the cognitive tasks that are present in sport. The high cognitive demands of the sporting environment therefore justify the inclusion of cognitive tasks in these return to sport tests. The aim of this research is to assess the impact of the cognitive task on the performance of a return to sport test following ACL reconstruction. Patients who have undergone ACL reconstruction and healthy subjects will therefore be given a return to sport test called the 'Single Leg Hop for Distance' with and without a cognitive task in order to observe the influence of the cognitive task on the results of the hop.

Including healthy subjects in this study will make it possible to study the impact of the cognitive task in these subjects, who have no neurophysiological dysfunction linked to ACL reconstruction.

The aim of this study is therefore to try to develop the return to sport tests currently described in the literature by proposing a new, improved test that takes account of the cognitive dimension, which is omnipresent in the sporting environment.

ELIGIBILITY:
The inclusion criteria for the test group (patients with ACL reconstruction) were as follows :

* Patients with an isolated, unilateral ACL rupture, corresponding to a first injury occurring without contact,
* Patients who have undergone surgical reconstruction using an autograft of the semitendinosus tendon alone, or an autograft of the semitendinosus tendon and gracilis, or BTB surgery,
* Patients at 6 +/- 1 months post-operative management,
* Patients aged between 16 and 40 included,
* Patients whose level of physical activity, assessed using the Tegner scale, is greater than or equal to 5.

Patients meeting all these inclusion criteria will be included in the study.

Thus, for the test group, the non-inclusion criteria to be taken into account are as follows:

* Patients with injuries associated with ACL rupture,
* Patients who have received conservative treatment or who have benefited from another surgical technique,
* Patients less than 5 months or more than 7 months post-operatively,
* Patients aged under 16 or over 40,
* Patients with a Tegner score of less than 5,
* Patients with recurrent homolateral or controlateral ACL rupture,
* Patients with an ACL rupture resulting from a direct or indirect impact injury mechanism.

Finally, for the test group, the exclusion criteria to be taken into account are as follows:

* Refusal to take part in the study,
* Withdrawal of the participant during the study,
* Loss of sight of the participant between the two weeks.

For the control group (healthy persons), the inclusion criteria are similar to those for the test group. They correspond to :

* Persons with no knee trauma in the six months prior to the start of the study,
* Persons between 16 and 40 years of age included,
* Persons whose level of physical activity, assessed using the Tegner scale, was greater than or equal to 5.

Persons meeting all these inclusion criteria will be included in the study.

Thus, for the control group, the non-inclusion criteria are as follows:

* Persons with knee lesions in the six months preceding the start of the study,
* Persons aged under 16 or over 40,
* Persons with a Tegner score strictly below 5.

Finally, the exclusion criteria for this group correspond to :

* Refusal to take part in the study,
* Retraction of the participant during the study,
* Loss of vision between the two weeks,
* Knee trauma between the two weeks.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Assessing the impact of the cognitive task on quantitative performance (jumping distance measured in meters) after ACL reconstruction. | 10 weeks
  Quantitative assessment of performance, using the Single Leg Hop for Distance, depending on whether or not a cognitive test is present.
  Measurement of jump distance in meters.

SECONDARY OUTCOMES:
Assessing the impact of the cognitive task on qualitative performance after ACL reconstruction with Qualitative Analysis of Single Leg Score. | 10 weeks
  Qualitative evaluation of the Single Leg Hop for Distance using Qualitative Analysis of Single Leg Score (QASLS), according to the presence or absence of a cognitive test.
  We use the Qualitative Analysis of Single Leg Score to evaluate the performance.
Assess the impact of the cognitive task on qualitative jumping performance after ACL reconstruction and in healthy subjects, with Qualitative Analysis of Single Leg Score. | 10 weeks
  Comparison of qualitative (Qualitative Analysis of Single Leg Score) jump performance between the two populations.
  We compare the Qualitative Analysis of Single Leg Score between the two population.
Assess the impact of the cognitive task on quantitative (distance measured in meters) jumping performance after ACL reconstruction and in healthy subjects. | 10 weeks
  Comparison of quantitative (distance in meters) jump performance between the two populations.
  We compare the jump distances measured in meters between the two populations.

CONTACTS AND LOCATIONS:
Overall Officials: Simon SV VALOT, Principal Investigator
Locations (4):
- France (4):
  - Orthosport Centre, Domont
  - Physiotherapy practice CESAL, Les Sables-d'Olonne
  - Institut de Formation en Masso-Kinésithérapie du Centre Hospitalier Universitaire de Poitiers (physiotherapy training institute), Poitiers
  - Physiotherapy practice MADINI, Poitiers

REFERENCES:
- [Background] Parry GN, Herrington LC, Munro AG. Reliability and Measurement Error of the Qualitative Analysis of Single Leg Loading (QASLS) Tool For Unilateral Tasks. Int J Sports Phys Ther. 2023 Oct 1;18(5):1136-1146. doi: 10.26603/001c.88007. eCollection 2023. PMID 37885771
- [Background] Li ZI, Green JS, Chalem I, Triana J, Rao N, Hughes AJ, Campbell KA, Jazrawi LM, Medvecky MJ, Alaia MJ. Patient-reported outcomes and return to pre-injury activities after surgical treatment of multi-ligamentous knee injuries in patients over 40-years-old: Average 5-years follow-up. Knee. 2024 Jan;46:89-98. doi: 10.1016/j.knee.2023.11.014. Epub 2023 Dec 8. PMID 38070381
- [Background] Hecker A, Schmaranzer F, Huber C, Maurer J, Egli RJ, Eberlein SC, Klenke FM. Treatment of Knee Dislocation With Primary Repair and Suture Augmentation: A Viable Solution. Orthop J Sports Med. 2022 Nov 17;10(11):23259671221132555. doi: 10.1177/23259671221132555. eCollection 2022 Nov. PMID 36425010
- [Background] Berk AN, Piasecki DP, Fleischli JE, Trofa DP, Saltzman BM. Trends in Patient-Reported Outcomes After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Orthop J Sports Med. 2023 May 31;11(5):23259671231174472. doi: 10.1177/23259671231174472. eCollection 2023 May. PMID 37284137
- [Background] Zhou W, Liu X, Hong Q, Wang J, Luo X. Association between passing return-to-sport testing and re-injury risk in patients after anterior cruciate ligament reconstruction surgery: a systematic review and meta-analysis. PeerJ. 2024 Apr 29;12:e17279. doi: 10.7717/peerj.17279. eCollection 2024. PMID 38699196
- [Background] Aizawa JY, Hirohata K, Ohji S, Mitomo S, Ohmi T, Koga H, Yagishita K. Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) subcategories are affected by subjective running ability and medial single-leg hop distance in postreconstruction patients at 6 months. J Exp Orthop. 2024 Feb 3;11(1):e12004. doi: 10.1002/jeo2.12004. eCollection 2024 Jan. PMID 38455451
- [Background] Measson MV, Ithurburn MP, Rambaud AJ. Intra-rater Reliability of a Qualitative Landing Scale for the Single-Hop Test: A Pilot Study. Int J Sports Phys Ther. 2022 Apr 1;17(3):493-500. doi: 10.26603/001c.33066. eCollection 2022. PMID 35391866
- [Background] Kiani Haft Lang M, Mofateh R, Orakifar N, Goharpey S. Differences in Neurocognitive Functions Between Healthy Controls and Anterior Cruciate Ligament-Reconstructed Male Athletes Who Passed or Failed Return to Sport Criteria: A Preliminary Study. J Sport Rehabil. 2023 Apr 25;32(6):645-654. doi: 10.1123/jsr.2022-0288. Print 2023 Aug 1. PMID 37185456
- [Background] Riera J, Forelli F, Coulondre C, Rambaud A. Fiche pratique du " Single Hop Test ". J Traumatol Sport. 1 mars 2023;40(1):46-8.
- [Background] Kotsifaki R, Korakakis V, King E, Barbosa O, Maree D, Pantouveris M, Bjerregaard A, Luomajoki J, Wilhelmsen J, Whiteley R. Aspetar clinical practice guideline on rehabilitation after anterior cruciate ligament reconstruction. Br J Sports Med. 2023 May;57(9):500-514. doi: 10.1136/bjsports-2022-106158. Epub 2023 Feb 2. PMID 36731908